CLINICAL TRIAL: NCT00290303
Title: Study to Show Non-inferiority of Tritanrix™-HepB/Hib-MenAC (+/- Hepatitis B Vaccine at Birth) Versus Tritanrix™-HepB/Hiberix™ Without Hepatitis B Vacc. at Birth for Antibody Response to All Vaccine Antigens Given in Healthy Infants
Brief Title: Assess if Immune Response of GSK Biologicals' Tritanrix™-HepB/Hib-MenAC Given Without or With Hepatitis B Vaccine at Birth is at Least as Good as Tritanrix™-HepB/Hiberix™ Without Hepatitis B Vaccine at Birth, When Given to Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 100478
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Haemophilus Influenzae Type b; Diphtheria; Whole Cell Pertussis; Hepatitis B; Tetanus
MeSH Terms: conditions — Haemophilus Infections; Diphtheria; Hepatitis B; Tetanus

INTERVENTIONS:
Biological: DTPw-HBV/Hib-MenAC conjugate vaccine

SUMMARY:
The purpose of this study is to compare the immune response, safety and reactogenicity of Tritanrix™-HepB/Hib-MenAC vaccine given either with or without a birth dose of hepatitis B vaccine to Tritanrix™-HepB/Hiberix™ when given to healthy infants (born to mothers who do not carry hepatitis B virus) at 6, 10 & 14 weeks of age. This study will also include a small group of infants born to mothers who do carry hepatitis B virus; these infants will receive a birth dose of hepatitis B vaccine and will be vaccinated with Tritanrix™ HepB/Hib-MenAC at 6, 10 & 14 weeks age.

DETAILED DESCRIPTION:
Randomized study with three groups (subjects born to mothers who do not carry hepatitis B virus) to receive one of the following vaccination regimens: - GSK Biologicals' Tritanrix™-HepB/Hib-MenAC and hepatitis B vaccine at birth

- GSK Biologicals' Tritanrix™-HepB/Hib-MenAC and no hepatitis B vaccine at birth - GSK Biologicals' Tritanrix™-HepB/Hiberix™ There will also be a fourth group (subjects born to mothers who do carry hepatitis B virus) to receive: - GSK Biologicals' Tritanrix™-HepB/Hib-MenAC and hepatitis B vaccine at birth

ELIGIBILITY:
Inclusion criteria:

* Healthy infants aged 3 days or less, written informed consent obtained from the parents, born after a gestation period of 36 to 42 weeks.
* Result of the maternal blood sample (presence/not of hepatitis B virus) is available.

Exclusion criteria:

* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period (except for immunoglobulins given at birth to infants born to HBsAg seropositive mothers).
* Acute disease at the time of enrolment.
* Known exposure to diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b and/or meningococcal disease.
* Hepatitis B vaccine given at birth outside the study.

Min Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 996 (Actual)
Dates: Start 2004-05; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: One month post-dose 3, measurement of serum bactericidal titers against meningococcal serogroups A & C (SBA-MenA; SBA-MenC), anti-PRP, anti-HBs & anti-diphtheria concentrations; & in some subjects anti-tetanus & anti-BPT concentrations.

SECONDARY OUTCOMES:
Reactogenicity and safety: After each vaccination, solicited (day 0-3, local & general) & unsolicited (day 0-30) symptoms. Over the full course of the study: serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Philippines (3):
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, Sampaloc, Manila

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 100478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 100478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 100478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 100478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 100478 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register